CLINICAL TRIAL: NCT03350542
Title: EVOLVE 48: A Prospective Multicenter Single Arm Trial to Assess the Safety and Effectiveness of the SYNERGY 48 mm Everolimus-Eluting Platinum Chromium Coronary Stent System for the Treatment of Atherosclerotic Lesion(s)
Brief Title: A Clinical Trial to Assess the SYNERGY 48 mm Stent System for the Treatment of Atherosclerotic Lesion(s)
Acronym: EVOLVE48
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2356
Record Dates: First submitted 2017-11-17; First posted 2017-11-22 (Actual); Results first posted 2021-02-05 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-04

CONDITIONS: Coronary Artery Disease
Keywords: Drug-Eluting Stents
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Prospective, open label, single arm, multi-center
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- SYNERGY 48 mm (Experimental): SYNERGY 48 mm is a device/ drug combination product composed of two components, a device (coronary stent system including a platinum chromium stent platform) and a drug product (a formulation of everolimus contained in a bioabsorbable polymer coating)
  Interventions: Device: SYNERGY 48 mm

INTERVENTIONS:
Device: SYNERGY 48 mm — A drug eluting coronary stent system

SUMMARY:
EVOLVE 48 is a prospective, open label, single arm, multi-center trial. The purpose of this study is to assess the FDA requirement for safety and effectiveness of the SYNERGY 48 mm Coronary Stent System for the treatment of subjects with atherosclerotic lesion(s) > 34 mm and ≤ 44 mm in length (by visual estimate) in native coronary arteries ≥2.5 mm to ≤4.0 mm in diameter (by visual estimate).

ELIGIBILITY:
Clinical Inclusion Criteria

* Subject must be at least 18 years of age
* Subject (or legal guardian) understands the trial requirements and the treatment procedures and provides written informed consent before any trial-specific tests or procedures are performed
* Subject is eligible for percutaneous coronary intervention (PCI) and is an acceptable candidate for coronary artery bypass grafting (CABG)
* Subject has either:

  * Symptomatic coronary artery disease with one of the following: stenosis ≥ 70%, abnormal fractional flow reserve (FFR), abnormal stress or imaging stress test, or elevated biomarkers prior to the procedure
  * OR
  * Documented silent ischemia based on one of the following: abnormal fractional flow reserve (FFR), abnormal stress or imaging stress test, or elevated biomarkers prior to the procedure
* Subject is willing to comply with all protocol-required follow-up evaluation Angiographic Inclusion Criteria (visual estimate)
* Target lesion must be located in a native coronary artery with a visually estimated reference vessel diameter (RVD) ≥2.5 mm and ≤4.0 mm
* Target lesion length must be >34 mm and ≤44 mm (by visual estimate)
* Target lesion must have visually estimated stenosis ≥50% and <100% with thrombolysis in Myocardial Infarction (TIMI) flow >1
* Coronary anatomy is likely to allow delivery of a study device to the target lesion
* The target lesion must be successfully predilated/pretreated. If a non-target lesion is treated, it should be treated first and should be deemed an angiographic success Note: Angiographic success is a mean lesion diameter stenosis < 50% (< 30% for stents) in 2 near-orthogonal projections with TIMI 3 flow, as visually assessed by the physician, without the occurrence of prolonged chest pain or ECG changes consistent with MI.

Note: Successful predilatation/pretreatment refers to dilatation with a balloon catheter of appropriate length and diameter, or pretreatment with directional or rotational coronary atherectomy, laser or cutting/scoring balloon with no greater than 50% residual stenosis and no dissection greater than National Heart, Lung, Blood Institute (NHLBI) type C.

Clinical Exclusion Criteria

* Subject has clinical symptoms and/or electrocardiogram (ECG) changes consistent with acute ST elevation MI (STEMI)
* Subject has cardiogenic shock, hemodynamic instability requiring inotropic or mechanical circulatory support, intractable ventricular arrhythmias, or ongoing intractable angina
* Subject has received an organ transplant or is on a waiting list for an organ transplant
* Subject is receiving or scheduled to receive chemotherapy within 30 days before or after the index procedure
* Planned PCI (including staged procedures) or CABG after the index procedure
* Subject previously treated at any time with intravascular brachytherapy
* Subject has a known allergy to contrast (that cannot be adequately premedicated) and/or the trial stent system or protocol-required concomitant medications (e.g., platinum, platinum-chromium alloy, stainless steel, everolimus or structurally related compounds, polymer or individual components, all P2Y12 inhibitors, or aspirin)
* Subject has one of the following (as assessed prior to enrollment):

  * Other serious medical illness (e.g., cancer, congestive heart failure) with estimated life expectancy of less than 24 months
  * Current problems with substance abuse (e.g., alcohol, cocaine, heroin, etc.)
  * Planned procedure that may cause non-compliance with the protocol or confound data interpretation
* Subject is receiving chronic (≥72 hours) anticoagulation therapy (i.e., heparin, coumadin) for indications other than acute coronary syndrome
* Subject has a platelet count <100,000 cells/mm3 or >700,000 cells/mm3
* Subject has a white blood cell (WBC) count < 3,000 cells/mm3
* Subject has documented or suspected liver disease, including laboratory evidence of hepatitis
* Subject is on dialysis or has baseline serum creatinine level >2.0 mg/dL (177µmol/L)
* Subject has a history of bleeding diathesis or coagulopathy or will refuse blood transfusions
* Subject has had a history of cerebrovascular accident (CVA) or transient ischemic attack (TIA) within the past 6 months
* Subject has an active peptic ulcer or active gastrointestinal (GI) bleeding
* Subject has signs or symptoms of active heart failure (i.e., New York Heart Association (NYHA) class IV) at the time of the index procedure
* Subject is participating in another investigational drug or device clinical trial that has not reached its primary endpoint
* Subject intends to participate in another investigational drug or device clinical trial within 12 months after the index procedure
* Subject with known intention to procreate within 12 months after the index procedure (women of child-bearing potential who are sexually active must agree to use a reliable method of contraception from the time of screening through 12 months after the index procedure)
* Subject is a woman who is pregnant or nursing Angiographic Exclusion Criteria (visual estimate)
* Subject has more than 1 target lesion, or more than 1 target lesion and 1 non-target lesion, which will be treated during the index procedure Note: Multiple focal stenoses will be considered as a single lesion if they can be completely covered with 1 study stent
* Treatment of lesions in more than 2 major epicardial vessels Note: 1 target lesion in the target vessel and 1 non-target lesion in non-target vessel is allowed
* Subject has unprotected left main coronary artery disease (>50% diameter stenosis)
* Subject has been treated with any type of PCI (i.e., balloon angioplasty, stent, cutting balloon atherectomy) within 24 hours prior to the index procedure
* Thrombus, or possible thrombus, present in the target vessel (by visual estimate)
* Target lesion meets any of the following criteria:
* Treatment of a single lesion with more than 1 stent
* Left main location
* Lesion is located within 3 mm of the origin of the left anterior descending (LAD) coronary artery or left circumflex (LCx) coronary artery by visual estimate
* Lesion is located within a saphenous vein graft or an arterial graft
* Lesion will be accessed via a saphenous vein graft or arterial graft
* Lesion with a TIMI flow 0 (total occlusion) or TIMI flow 1 prior to guide wire crossing
* Lesion treated during the index procedure that involves a complex bifurcation (e.g., bifurcation lesion requiring treatment with more than 1 stent)
* Lesion is restenotic from a previous stent implantation or study stent would overlap with a previous stent
* Non-target lesion meets any of the following criteria:
* Located within the target vessel
* Left main location
* Lesion is located within a saphenous vein graft or an arterial graft
* Lesion with a TIMI flow 0 (total occlusion) or TIMI flow 1 prior to guide wire crossing
* Lesion treated during the index procedure that involves a complex bifurcation (e.g., bifurcation lesion requiring treatment with more than 1 stent)
* Requires additional unplanned stents (treatment of the non-target lesion with more than one stent is permitted as long as the stents are initially planned)
* Treatment not deemed an angiographic success Note: Angiographic success is a mean lesion diameter stenosis < 50% (< 30% for stents) in 2 near-orthogonal projections with TIMI 3 flow, as visually assessed by the physician, without the occurrence of prolonged chest pain or ECG changes consistent with MI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2020-01-16 (Actual); Study Completion 2021-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Karmpaliotis, MD, Principal Investigator — New York Presbyterian Hospital
Locations (15):
- United States (8):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - HealthEast St. Joseph's Hospital, Saint Paul, Minnesota
  - New York Presbyterian Hospital - Columbia University Medical Center, New York, New York
  - Rex Hospital, Raleigh, North Carolina
  - Lindner Center for Research and Education at Christ Hospital, Cincinnati, Ohio
  - York Hospital, York, Pennsylvania
  - Baylor Heart & Vascular Hospital, Dallas, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
- P. Stradins University Hospital, Riga, Latvia
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - North Shore Hospital, Takapuna
- United Kingdom (4):
  - Royal Victoria Hospital, Belfast
  - Golden Jubilee National Hospital, Glasgow
  - Freeman Hospital, Newcastle upon Tyne
  - John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 100 patients have been enrolled in the study from April 12, 2018 until January 17, 2019. The Evolve 48 study is anticipated to be completed (final 2-year follow up) in 2021.
Period: Overall Study
Arm/Group | SYNERGY 48 mm
Started | 100
Completed 12-Month Clinical F/U | 96
Death With no 12-month F/U | 4
Completed | 96
Not Completed | 4

BASELINE CHARACTERISTICS:
Groups:
- SYNERGY 48mm: SYNERGY is a device/drug combination product comprised of two regulated components: a device (Coronary Stent System) and a drug product (a formulation of everolimus contained in a bioabsorbable polymer coating).
Arm/Group | SYNERGY 48mm
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.99 (10.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 60
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska native | 0
  Black, of African heritage | 6
  Caucasian | 85
  Hispanic | 3
  Native Hawaiian or other Pacific Islander | 1
  Other | 5
  Not disclosed | 0
Region of Enrollment [Number; unit: participants]
  New Zealand | 19
  Latvia | 3
  United States | 45
  United Kingdom | 33
Smoking [Count of Participants; unit: Participants]
  Smoking, ever | 51
  Smoking, current | 14
  Smoking, previous | 37
Medically Treated Diabetes [Count of Participants; unit: Participants] | 27
Hyperlipidemia requiring medication [Count of Participants; unit: Participants] | 82
Hypertension requiring medication [Count of Participants; unit: Participants] | 76
History of bleeding disorder [Count of Participants; unit: Participants] | 4
History of Transient Ischemic Attack (TIA) or Coronary vasospasm (CVA) [Count of Participants; unit: Participants] — Population: For baseline categorical variables, "unknown" responses and missing values will not be counted in rate denominators
  Participants
    number analyzed (Participants) | 99
    (all) | 4
History of TIA [Count of Participants; unit: Participants] — Population: For baseline categorical variables, "unknown" responses and missing values will not be counted in rate denominators
  Participants
    number analyzed (Participants) | 98
    (all) | 4
History of CVA [Count of Participants; unit: Participants] — Population: For baseline categorical variables, "unknown" responses and missing values will not be counted in rate denominators
  Participants
    number analyzed (Participants) | 99
    (all) | 0
History of renal disease [Count of Participants; unit: Participants] | 10
History of Peripheral Vascular Disease (PVD) [Count of Participants; unit: Participants] — Population: For baseline categorical variables, "unknown" responses and missing values will not be counted in rate denominators
  Participants
    number analyzed (Participants) | 99
    (all) | 10
Baseline lesion characteristics as determined by the Angiographic core lab, ITT analysis set [Count of Participants; unit: Participants] — Intent-to-Treat (ITT)
  Participants
    Left Anterior Descending (LAD) | 40
    Left Circumflex Artery (LCx) | 14
    Right Coronary Artery (RCA) | 46
    Left Main Coronary Artery (LMCA) | 0

OUTCOME MEASURES:

1. Primary Outcome: Target Lesion Failure Rate at 12-months
Description: The primary endpoint is the 12-month Target Lesion Failure (TLF) rate, defined as any ischemia-driven revascularization of the target lesion (TLR), myocardial infarction (MI, Q-wave and non-Q-wave) related to the target vessel, or cardiac death.
Time Frame: 12-month
Population: The per-protocol and ITT populations are the same.
Measure: Number; unit: percentage of participants
Arm/Group | SYNERGY 48 mm
Number analyzed (Participants) | 98
percentage of participants | 4

2. Secondary Outcome: Target Lesion Revascularization (TLR) Rate at 12 Months
Description: The TLR overall rate includes: TLR Percutaneous Coronary Intervention (PCI) and TLR Coronary Artery Bypass Graft (CABG)
Time Frame: 12 months
Population: Intent-to-Treat population
Measure: Number; unit: percentage of participants
Arm/Group | SYNERGY 48 mm
Number analyzed (Participants) | 100
percentage of participants | 1

3. Secondary Outcome: Target Vessel Revascularization (TVR) Rate at 12 Months.
Description: TVR overall includes: TVR PCI and TVR CABG
Time Frame: 12 months
Population: Intent-to-Treat
Measure: Number; unit: percentage of participants
Arm/Group | SYNERGY 48 mm
Number analyzed (Participants) | 100
percentage of participants | 1

4. Secondary Outcome: Target Vessel Failure (TVF) Rate at 12 Months
Description: Target Vessel Failure is defined as any ischemic-driven revascularization of the target vessel, MI related to the target vessel, or any cardiac death.
Time Frame: 12 months
Population: Intent-to-Treat analysis
Measure: Number; unit: percentage of participants
Arm/Group | SYNERGY 48 mm
Number analyzed (Participants) | 100
percentage of participants | 4

5. Secondary Outcome: MI (Q-wave and Non-Q-wave) Rate
Description: The MI rate includes: MIs related to the Target Vessel, MIs with unknown relationship to the Target Vessel and MIs not related to the Target Vessel.
Time Frame: 12 months
Population: Intent-to-Treat analysis
Measure: Number; unit: percentage of participants
Arm/Group | SYNERGY 48 mm
Number analyzed (Participants) | 100
percentage of participants | 2

6. Secondary Outcome: Cardiac Death Rate
Description: Cardiac death is defined as death due to any of the following; acute MI, cardiac perforation/pericardial tamponade, arrhythmia or conduction abnormality, CVA through hospital discharge or CVA suspected of being related to the procedure, death due to complication of the procedure, including bleeding, vascular repair, transfusion reaction, or bypass surgery and any death in which a cardiac cause cannot be excluded.
Time Frame: 12 months
Population: Intent-to-Treat
Measure: Number; unit: percentage of participants
Arm/Group | SYNERGY 48 mm
Number analyzed (Participants) | 100
percentage of participants | 1

7. Secondary Outcome: Non-cardiac Death Rate
Description: Non-cardiac death is defined as a death not due to cardiac causes as previously defined.
Time Frame: 12 months
Measure: Number; unit: percentage of participants
Arm/Group | SYNERGY 48 mm
Number analyzed (Participants) | 100
percentage of participants | 4

8. Secondary Outcome: All Death Rate
Time Frame: 12 months
Measure: Number; unit: percentage of participants
Arm/Group | SYNERGY 48 mm
Number analyzed (Participants) | 100
percentage of participants | 5

9. Secondary Outcome: Cardiac Death or MI Rate
Time Frame: 12 months
Measure: Number; unit: percentage of participants
Arm/Group | SYNERGY 48 mm
Number analyzed (Participants) | 100
percentage of participants | 3

10. Secondary Outcome: All Death or MI Rate
Time Frame: 12 months
Population: Intent-to-Treat
Measure: Number; unit: percentage of participants
Arm/Group | SYNERGY 48 mm
Number analyzed (Participants) | 100
percentage of participants | 6

11. Secondary Outcome: All Death/MI/TVR Rate
Time Frame: 12 months
Measure: Number; unit: percentage of participants
Arm/Group | SYNERGY 48 mm
Number analyzed (Participants) | 100
percentage of participants | 7

12. Secondary Outcome: Stent Thrombosis Rate
Time Frame: 12 months
Population: Intent-to-Treat
Measure: Number; unit: percentage of participants
Arm/Group | SYNERGY 48 mm
Number analyzed (Participants) | 100
percentage of participants | 0

13. Secondary Outcome: Periprocedural Technical Success Rate
Description: Successful delivery and deployment of the study stent to the target vessel, without balloon rupture or stent embolization, and post-procedure diameter stenosis of <30% in 2 near-orthogonal projections with Thrombolysis in Myocardial Infarction (TIMI) 3 flow in the target lesion, as visually assessed by the physician.
Time Frame: Day 1 (periprocedural)
Population: Intent-to-Treat
Measure: Number; unit: percentage of participants
Arm/Group | SYNERGY 48 mm
Number analyzed (Participants) | 100
percentage of participants | 100

14. Secondary Outcome: Periprocedural Clinical Procedural Success Rate
Description: Post-procedure lesion diameter stenosis <30% in 2 near-orthogonal projections with TIMI 3 flow in the target lesion, as visually assessed by the physician, without the occurrence of in-hospital cardiac death, MI, or TVR.
Time Frame: 12 months
Population: Intent-to-Treat
Measure: Number; unit: percentage of participants
Arm/Group | SYNERGY 48 mm
Number analyzed (Participants) | 100
percentage of participants | 100

ADVERSE EVENTS:
Time Frame: Site-Reported Serious Adverse Events (SAE) to 12 Months
Description: For All Cause Mortality, the at risk population (denominator) is the ITT population.
  For the SAE/AE tables, the at risk population (denominator) is the ITT population.
Arm/Group | SYNERGY 48 mm
All-Cause Mortality (participants affected / at risk) | 5/100
Serious Adverse Events (participants affected / at risk) | 31/100
Other Adverse Events (participants affected / at risk) | 4/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SYNERGY 48 mm (N=100)
Coronary artery dissection (Cardiac disorders) | 8
Plaque shift (Injury, poisoning and procedural complications) | 3
Colitis (Gastrointestinal disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 4
Carotid artery stenosis (Nervous system disorders) | 2
Osteomyelitis (Infections and infestations) | 1
Intermittent claudication (Vascular disorders) | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 1
Fluid overload (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anxiety (Psychiatric disorders) | 1
Angina pectoris (Cardiac disorders) | 4
Acute coronary syndrome (Cardiac disorders) | 2
Cardiac failure congestive (Cardiac disorders) | 2
Acute myocardial infarction (Cardiac disorders) | 1
Angina unstable (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiogenic shock (Cardiac disorders) | 1
Cardiomyopathy (Cardiac disorders) | 1
Chronic left ventricular failure (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Coronary artery stenosis (Cardiac disorders) | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1
Intentional overdose (Injury, poisoning and procedural complications) | 1
Postoperative wound complication (Injury, poisoning and procedural complications) | 1
Colitis ischaemic (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Cellulitis (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Orthostatic hypotension (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1
Peripheral ischaemia (Vascular disorders) | 1
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SYNERGY 48 mm (N=100)
Angina unstable (Cardiac disorders) | 1
Blood creatine phosphokinase MB increased (Investigations) | 1
Coronary artery occlusion (Cardiac disorders) | 1
Electrocardiogram T wave abnormal (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A contractual agreement is in place between the PI and the Sponsor that restricts the rights to discuss or publish trial results without prior review by the sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-16): https://cdn.clinicaltrials.gov/large-docs/42/NCT03350542/Prot_SAP_000.pdf